CLINICAL TRIAL: NCT03472365
Title: A Randomized Phase 2 Study to Evaluate Safety and Efficacy of the Combination of SHR-1210 With Capecitabine + Oxaliplatin or Apatinib as First-line Treatment in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of SHR-1210 in Combination With Capecitabine + Oxaliplatin or Apatinib in Treatment of Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-207
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: PD-1; SHR-1210; Capecitabine; Oxaliplatin; Apatinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Capecitabine; Oxaliplatin; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants receive SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus capecitabine 1000 mg/m^2 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days, plus oxaliplatin 130 mg/m^2, IV q3w; for 4-6 cycles followed by SHR-1210 plus apatinib 375 mg PO qd if there is no PD.
  Interventions: Biological: SHR-1210; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Apatinib
- Cohort 2 (Experimental): Participants receive SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus apatinib 375 mg daily (QD) continuous oral administration of each 3-week cycle.
  Interventions: Biological: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody
  Other Names: Camrelizumab
Drug: Capecitabine — 1000 mg/m^2 administered as continuous oral twice daily (BID) of each 3-week cycle.
  Arms: Cohort 1
Drug: Oxaliplatin — 130 mg/m^2 administered IV Q3W on Day 1 of each 3-week cycle.
  Arms: Cohort 1
Drug: Apatinib — 375 mg administered as continuous oral once daily (QD) of each 3-week cycle.

SUMMARY:
The purpose of this trial is to estimate overall response rate (ORR) of SHR-1210 combined with capecitabine and oxaliplatin or with apatinib as first-line treatment in subjects with locally advanced or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
Approximately 110 participants will be assigned to SHR-1210 + capecitabine + oxaliplatin combination therapy (Cohort 1), or SHR-1210 + apatinib combination therapy (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic adenocarcinoma of stomach or the esophagogastric junction (GEJ).
* Age ≥ 18 years old, male or female.
* NO previous therapy for advanced/metastatic disease of GC/GEJ (including HER2 inhibitor). Subjects with previous adjuvant/neo-adjuvant therapy completed more than 6 months can be enrolled.
* Has measurable disease per RECIST 1.1.
* Life expectancy ≥ 12 weeks.
* Eastern Cooperative Group (ECOG) performance status of 0 to 1.
* Has adequate organ function.
* Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and must not be pregnant or breast-feeding women. If the result is negative, she must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs. And non-sterilized males who are sexually active must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs.

Exclusion Criteria:

* Has known HER2-positive status.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, or a VEGFR inhibitor.
* Has known active central nervous system metastases.
* Has received a live vaccine within 4 weeks prior to the first dose of study treatment.
* With any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention.
* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
* Coagulation abnormalities (INR > 1.5 or APTT > 1.5×ULN), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng Z, Wei J, Wang F, Ying J, Deng Y, Gu K, Cheng Y, Yuan X, Xiao J, Tai Y, Wang L, Zou J, Zhang Y, Shen L. Camrelizumab Combined with Chemotherapy Followed by Camrelizumab plus Apatinib as First-line Therapy for Advanced Gastric or Gastroesophageal Junction Adenocarcinoma. Clin Cancer Res. 2021 Jun 1;27(11):3069-3078. doi: 10.1158/1078-0432.CCR-20-4691. Epub 2021 Mar 25. PMID 33766817

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants received SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus capecitabine 1000 mg/m^2 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days, plus oxaliplatin 130 mg/m^2, IV q3w; for 4-6 cycles followed by SHR-1210 plus apatinib 375 mg PO qd if there was no PD.
- Cohort 2: Participants received SHR-1210 200 mg, intravenously (IV) every 3 weeks(Q3W) plus apatinib 375 mg daily (QD) continuous oral administration of each 3-week cycle.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 48 | 19
Completed | 48 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 48 | 19 | 67
Age, Continuous [Median (Full Range); unit: Years old] | 56.0 [23 to 73] | 62.0 [27 to 72] | 59.0 [23 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 16 | 53
  Male | 11 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 48 | 19 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 48 | 19 | 67

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Time Frame: Up to approximately 6 months.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 48 | 19
percentage | 58.3 [43.2 to 72.4] | 10.5 [1.3 to 33.1]

2. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
Time Frame: Up to 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 48 | 19
months | 6.768 [5.552 to 9.495] | 2.793 [1.380 to 4.764]

3. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: For participants who demonstrate CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), DOR is defined as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1 based on assessments by blinded independent central review or death due to any cause, whichever occurs first.
Time Frame: Up to 24 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 48 | 19
months | 5.749 [4.370 to 8.345] | NA [2.694 to NA] — The median DoR was not reached.

4. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1
Description: DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1.
Time Frame: Up to 24 months.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 48 | 19
percentage | 93.8 [82.8 to 98.7] | 57.9 [33.5 to 79.7]

5. Secondary Outcome: Number of Subjects With Treatment-related Adverse Events (AEs)
Description: Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
Time Frame: Up to 24 months.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 48 | 19
participants | 48 | 18

ADVERSE EVENTS:
Time Frame: 32 months
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 14/48 | 9/19
Serious Adverse Events (participants affected / at risk) | 22/48 | 12/19
Other Adverse Events (participants affected / at risk) | 48/48 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=48) | Cohort 2 (N=19)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Platelet count decreased (Investigations) | 5 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Liver injury (Hepatobiliary disorders) | 0 | 2
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=48) | Cohort 2 (N=19)
Anaemia (Blood and lymphatic system disorders) | 24 | 9
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 0
Hypothyroidism (Endocrine disorders) | 8 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 24 | 5
Vomiting (Gastrointestinal disorders) | 18 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 3
Abdominal distension (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 18 | 4
Pyrexia (General disorders) | 15 | 8
Pain (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 4
Liver injury (Hepatobiliary disorders) | 1 | 1
Reactive capillary endothelial proliferation (Immune system disorders) | 38 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 32 | 4
Neutrophil count decreased (Investigations) | 30 | 7
White blood cell count decreased (Investigations) | 26 | 7
Aspartate aminotransferase increased (Investigations) | 21 | 6
Alanine aminotransferase increased (Investigations) | 16 | 9
Gamma-glutamyltransferase increased (Investigations) | 15 | 8
Weight decreased (Investigations) | 14 | 8
Bilirubin conjugated increased (Investigations) | 12 | 4
Blood bilirubin increased (Investigations) | 12 | 5
Blood alkaline phosphatase increased (Investigations) | 11 | 4
Blood thyroid stimulating hormone increased (Investigations) | 11 | 2
Blood creatine phosphokinase increased (Investigations) | 7 | 3
Blood lactate dehydrogenase increased (Investigations) | 7 | 2
Blood bilirubin unconjugated increased (Investigations) | 6 | 0
Occult blood positive (Investigations) | 5 | 4
Weight increased (Investigations) | 5 | 0
Electrocardiogram QT prolonged (Investigations) | 4 | 0
Blood creatine phosphokinase MB increased (Investigations) | 3 | 2
Blood urea increased (Investigations) | 3 | 0
Fibrin D dimer increased (Investigations) | 3 | 2
Protein urine present (Investigations) | 3 | 2
Tri-iodothyronine decreased (Investigations) | 3 | 0
Tri-iodothyronine free decreased (Investigations) | 3 | 2
Urine output decreased (Investigations) | 3 | 0
White blood cell count increased (Investigations) | 3 | 0
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 2 | 2
C-reactive protein increased (Investigations) | 2 | 1
Blood cholinesterase decreased (Investigations) | 1 | 1
Thyroxine free decreased (Investigations) | 1 | 1
Urine ketone body present (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Anti-thyroid antibody positive (Investigations) | 0 | 1
Bilirubin urine present (Investigations) | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 1
Coagulation test abnormal (Investigations) | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Urine bilirubin increased (Investigations) | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 6
Decreased appetite (Metabolism and nutrition disorders) | 11 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 5 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 19 | 0
Neurotoxicity (Nervous system disorders) | 6 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 5 | 1
Proteinuria (Renal and urinary disorders) | 16 | 5
Haematuria (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 11 | 6
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03472365/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03472365/SAP_001.pdf